MCC-15-11083 NCT02957968

T-Cell Immune Checkpoint Inhibition Plus Hypomethylation for Locally Advanced HER2-Negative Breast Cancer - A Phase 2 Neoadjuvant Window Trial of Pembrolizumab and Decitabine Followed by Standard Neoadjuvant Chemotherapy

10/12/2022

## RESEARCH PARTICIPANT INFORMED CONSENT FORM

**TITLE:** T-Cell Immune Checkpoint Inhibition Plus Hypomethylation for Locally

Advanced HER2-Negative Breast Cancer – A Phase 2 Neoadjuvant Window Trial of Pembrolizumab and Decitabine Followed by Standard Neoadjuvant

Chemotherapy

**PROTOCOL #:** MCC-15-11083

**VCU IRB #**: HM20008607

**SPONSOR-** Harry D. Bear, MD, PhD

**INVESTIGATOR:** Virginia Commonwealth University (VCU)

Massey Cancer Center Box 980011, VCUHS Richmond, VA 23298-0011

804-828-9325

### INTRODUCTION

This consent form will tell you about this research study, which is also called a clinical trial. Your study doctor or study team will explain the research study to you. Research studies only include people who choose to take part. You have the option to not participate. You may take home an unsigned copy of this consent form so that you can discuss the study with your family or friends before making your decision. You may also discuss it with your health care team. If you have any questions, ask your study doctor or study team for more explanation. Please take your time to make your decision about taking part in this study.

### OVERVIEW AND KEY INFORMATION

### Taking part in this study is your choice

You can choose to take part or you can choose not to take part in this study. You also can change your mind at any time. Whatever choice you make, you will not lose access to your medical care or give up any legal rights or benefits.

## What is the usual approach to treating my cancer?

You are being asked to take part in this study because you have locally advanced HER2-negative breast cancer. Your doctors have determined that the right treatment approach for you is to receive chemotherapy before surgery to shrink the tumor so that surgery can be performed with a better outcome. Treatment given before surgery is called "neoadjuvant therapy." Radiation therapy may be given after surgery or instead of surgery, if breast surgery is not possible. If the cancer has estrogen or progesterone receptors, treatment with drugs called endocrine therapy are also a part of the usual approach when treating locally advanced breast cancer.

## Why is this study being done?

Activation of the immune system is an important part of the body's response to try to get rid of cancer cells. Cancers are able to develop and may grow more rapidly when the immune system is not able to get rid of cancer cells. Testing in clinical trials has shown that breast cancers with evidence of a partial immune response have a better response to neoadjuvant chemotherapy and a greater chance of a complete response. A complete response means that cancer cells were killed by neoadjuvant chemotherapy, and no remaining cancer was found at the time of surgery. Patients who have a complete response to neoadjuvant chemotherapy have the highest rates of cure from neoadjuvant chemotherapy. Researchers are hoping to increase the chance of a complete response to neoadjuvant chemotherapy by finding ways to improve the immune response to breast cancer.

The purpose of this study is to test if a short course of immunotherapy with 2 study drugs, decitabine given daily for 4 days followed by 2 doses of pembrolizumab given 2 weeks apart, before standard neoadjuvant chemotherapy begins will improve the immune response in the cancer and increase how often a complete response occurs with standard chemotherapy. The study will also look for side effects caused by the immunotherapy. Laboratory tests have shown that the combination of decitabine followed by pembrolizumab may increase immune response in and around the tumor. The study drugs may also be able to change tumor cells in ways that improve the benefit of standard neoadjuvant chemotherapy.

Decitabine has been approved by the Food and Drug Administration (FDA) for treatment of myelodysplastic syndromes, which are cancers involving blood cells and bone marrow. Pembrolizumab has been approved by the FDA for the treatment of a number of different cancer types including advanced melanoma and some types of advanced triple negative breast cancer whose tumors express PD-L1 as determined by an FDA-approved test, lung cancer, head and neck cancer, and esophageal cancer. Decitabine and pembrolizumab have not been approved by the FDA for treatment of breast cancer before surgery and are experimental in this study.

Dr Bear, the sponsor-investigator for this study, has a paid consulting relationship with Merck & Company. Merck is supporting this study and providing the pembrolizumab.

There will be up to 50 participants in this study. Participants will be enrolled at the VCU Massey Cancer Center and other cancer centers in the United States.

## What are the risks and benefits of taking part in this study?

There are both risks and benefits to taking part in this study. It is important for you to think carefully about these as you make your decision. We want you to know about a few key risks right now. We will give you more information in the "WHAT POSSIBLE RISKS CAN I EXPECT FROM TAKING PART IN THIS STUDY?" section.

## Risks

We want to make sure you know about a few key risks right now. We give you more information in the "What possible risks can I expect from taking part in this study?" section.

If you choose to take part in this study, there is a risk that decitabine and pembrolizumab may not be as good as other drugs at shrinking or stabilizing your cancer.

There is also a risk that you could have side effects from the decitabine and pembrolizumab. These side effects may be worse and may be different than you would get with the usual approach for your cancer.

Some of the most common side effects that the study doctors know about are:

- Decreased numbers of some types of blood cells
- Nausea
- Vomiting
- Allergic reaction
- Inflammation of any organ or body system

### **Benefits**

It is not possible to know at this time if the study approach of adding immunotherapy before standard neoadjuvant chemotherapy will be effective in bringing about changes in the tumor that will improve the benefits of neoadjuvant chemotherapy. It is unlikely that the combination of decitabine and pembrolizumab will help you live longer. This study may help the study doctors learn things that may help other people in the future.

## What are my other choices if I do not take part in this study?

If you decide not to take part in this study, you have other choices. For example:

- You may choose to have chemotherapy before surgery without being in a research study.
- If it is possible to have breast surgery without neoadjuvant therapy, you may choose to have chemotherapy and other types of treatment after surgery.
- You may choose to take part in a different study, if one is available.
- Or you may choose not to be treated.

Now that you have a general overview of the study, we want to provide the details about what your participation involves. Please read, or have someone read to you, the rest of this document. If there is anything you don't understand, be sure to ask your study doctor or study team.

### HOW WILL MY CANCER BE TREATED IF I TAKE PART IN THIS STUDY?

All study participants will receive 2 immunotherapy study drugs followed by standard neoadjuvant chemotherapy for locally advanced breast cancer. Surgery, if possible, will be performed after completion of the neoadjuvant chemotherapy.

Immunotherapy Study Treatment

You will first be given 2 immunotherapy study drugs. Both drugs will be given to you at the Massey Cancer Center.

- Decitabine will be given into a vein (IV) once daily for 4 days
- After completing decitabine, pembrolizumab will be given IV with the second treatment given about 2 weeks later

## Standard Neoadjuvant Chemotherapy

You will then receive standard chemotherapy which can be given to you at the Massey Cancer Center or by your medical oncologist at a Massey Cancer Center Affiliate Network center.

- Doxorubicin and cyclophosphamide (AC) will be given IV every 2 or 3 weeks for 4 treatments
- Paclitaxel or Nab-paclitaxel will be given IV every week for 12 weeks after completing AC.
   If you are not one of the first 11 patients in this study, your medical oncologist may decide to give you paclitaxel or Nab-paclitaxel first and then AC.
- If you have triple negative breast cancer (a type of breast cancer that does **not** have HER2, estrogen, or progesterone receptors), carboplatin will be given IV every week or every 3 weeks, with paclitaxel or Nab-paclitaxel every week, for 12 weeks.

### Surgery

After completing all neoadjuvant therapy, breast surgery and evaluation of nearby lymph nodes will be performed. Your surgery can be performed by a breast surgeon at Massey Cancer Center or by your community breast surgeon.

The chart below shows the treatment included in the study. Start reading at the left side and read across to the right, following the arrows.



### Extended Pembrolizumab Treatment

If you have triple negative breast cancer, your study doctor may discuss the option of additional pembrolizumab treatments. Pembrolizumab may be included with standard neoadjuvant chemotherapy and given after surgery because initial clinical trials suggest that this may be more effective at treating your type of cancer. If your study doctor agrees this is the best choice for you, you will be given pembrolizumab treatments IV every 3 weeks during standard neoadjuvant chemotherapy, 4 treatments over 12 weeks. Starting 1 or 2 months after your surgery, you will be given pembrolizumab treatments IV every 3 weeks, up to 8 treatments.

### **HOW LONG WILL I BE IN THIS STUDY?**

You will be in this study for up to about 18 months, or a year and a half. Your study doctor will check on the status of your cancer and whether you have had any side effects for about a month after you have surgery. If you do not have surgery, your study doctor will check on the status of your cancer and watch for side effects for about a month after the decision not to have surgery. About 1 year after surgery (or the decision not to have surgery), your doctor will check your disease status and if you have had any new pembrolizumab side effects. If you had pembrolizumab side effects during treatment or during the month or so after treatment, your doctor will also check on the status of those side effects.

### WHAT EXTRA TESTS AND PROCEDURES WILL I HAVE IF I TAKE PART IN THIS STUDY?

If you plan to have treatment for your breast cancer and decide to take part in this study, most of the exams, tests, and procedures you will have are the usual approach in treating HER2-negative locally advanced breast cancer before having surgery. Your study doctor or study team will tell you about these.

To check for any side effects of the immunotherapy study drugs, extra blood tests and physical exams will be performed after the last decitabine treatment and after the last pembrolizumab treatment before chemotherapy.

This study also includes research using tumor and blood samples to learn about the immune response to study treatment in the tumor cells.

This study does not plan to use your samples to sequence all or part of your DNA. If any inventions or discoveries result from the use of your samples, there are no plans to share any money or profits with you.

### Biopsies to Collect Tumor Samples for Research Purposes

If you take part in this study, you will need to have a needle biopsy to remove 4 samples of tumor at each of 2 time points during the study to collect tumor samples for research purposes. The biopsies are required in this study because the research using the tumor samples is one of the main purposes of the study. You will have the needle biopsies at the following times:

- Before the first decitabine treatment
- After the last pembrolizumab treatment before chemotherapy

Common side effects of a needle biopsy are a small amount of bleeding at the time of the procedure, pain at the biopsy site, which can be treated with regular pain medications, and bruising. Rarely, an infection or more serious bleeding may occur.

### Collection of Tumor Samples Removed at the time of Surgery

If you have breast surgery, your study doctor will obtain samples of tumor or nearby breast tissue that was removed during your breast surgery.

### Tumor Samples for Research Purposes

Your tumor samples will be used to look for and evaluate lymphocytes and other immune system cells in and around your tumor. Your tumor samples will also be tested for molecular features of the immune system cells and their response to treatment. Some tests using part of

your tumor sample will be performed by Merck & Company. Tumor samples will continue to be used until they are used up.

Tests using your tumor sample will not be done for any routine clinical use and they cannot determine if you have a gene mutation that can be passed on in families. The results will not be added to your medical record and you and your study doctor will not know the results.

Results from the research will be placed in a storage system called a database. Some of the molecular information and your health information may be placed in the database. The database will not include your name or other personal identifying information. Data in the database may be accessed only by approved researchers.

## Blood Samples for Research Purposes

This study also includes research using blood samples to study the effects of the study drugs on immune system cells found in the blood. These blood samples are required in this study because the research on the sample is an important part of the study. Blood samples each measuring about a teaspoon will be collected at the following times:

- Before beginning the study treatment
- After the last decitabine treatment
- After the last pembrolizumab treatment before chemotherapy

Common side effects of blood sample collection are brief pain and bleeding or bruising at the puncture site used to collect the blood sample. There is also a small risk of infection, light-headedness, and fainting.

The results of the research using your blood samples will not be provided to you. The samples are collected only for the research study. There will be no benefit to you.

### WHAT POSSIBLE RISKS CAN I EXPECT FROM TAKING PART IN THIS STUDY?

The drugs used in this study may affect how different parts of your body work for example your liver and blood. The study doctor will be testing your blood and will let you know if changes occur that may affect your health.

Here are important points about side effects:

- Your study doctor does not know who will or will not have side effects
- Some side effects may go away soon, some may last a long time, or some may never go away
- Some side effects may interfere with your ability to have children
- Some side effects may be serious, may even result in death, and may occur after study treatment has ended

Here are important points about how you and your study doctor can make side effects less of a problem:

 Tell your study doctor or study team if you notice or feel anything different so they can see if you are having a side effect

- Your study doctor may be able to treat some side effects
- Your study doctor may adjust the drugs to try to reduce side effects

The tables on the next pages show the most common and the most serious side effects that researchers know about. The side effects listed for decitabine were reported in research studies evaluating ongoing treatment for myelodysplastic syndromes. The side effects listed for pembrolizumab were reported in research studies evaluating ongoing treatment for advanced melanoma and lung cancer. The side effects listed for the standard neoadjuvant chemotherapy drugs (doxorubicin, cyclophosphamide, paclitaxel, Nab-paclitaxel, and carboplatin) have been reported during extensive use of these drugs to treat breast and other types of cancer.

Researchers do not yet know whether the side effects listed on the table will occur more often or be worse when immunotherapy is given before chemotherapy. If important new information is learned about side effects, your study doctor will discuss these with you.

Let your study doctor or study team know of any questions you have about possible side effects. You can ask your study doctor questions about side effects at any time.

### **Known Side Effects of Decitabine**

### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving **decitabine**, more than 20 may have:

- Low number of white blood cells which could increase the chance of having an infection
- Low number of platelets in the blood which may cause bleeding and bruising
- Anemia, which may cause tiredness and may require transfusion
- Fever
- Constipation
- Diarrhea
- Nausea and loss of appetite
- Tiredness
- Swelling of hands and feet
- Shortness of breath and cough
- Headache
- Dizziness

### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving **decitabine**, from 4 to 20 may have:

- Sores in the mouth and esophagus which may be painful and cause difficulty swallowing
- Indigestion, vomiting, and abdominal pain
- Dehydration
- Infection
- Chills
- Weight loss
- Pain including chest, ear, back, and other bones
- Muscle aches and spasms
- Increase or decrease in blood pressure
- Skin changes including rash, itchiness, redness, and dryness
- Heart failure
- Rapid heart beats
- Chest pain
- Collection of fluid around the lungs in the chest cavity
- Difficulty sleeping
- Night sweats
- Anxiety, depression, and confusion
- Decrease in levels of potassium and magnesium in the blood
- Increase in blood sugar
- Increase in bilirubin in the blood, a liver test indicating possible liver damage

### RARE, AND SERIOUS

In 100 people receiving **decitabine**, 3 or fewer may have:

- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Changes in heart rhythm and heart attack
- Kidney failure

### **Known Side Effects of Pembrolizumab**

Pembrolizumab works by helping your immune system to fight your cancer.

However, pembrolizumab can also cause your immune system to attack normal organs and tissues in your body and can affect the way they work, which can result in side effects. These side effects may be serious (i.e., causing hospitalization or be life-threatening), may result in death, and/or may occur after you stop taking pembrolizumab. These side effects can affect more than one of your normal organs and tissues at the same time.

## **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving **pembrolizumab**, 20 or more may have:

- Itching of the skin
- · Loose or watery stools
- Cough

### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving **pembrolizumab**, from 5 to 19 may have:

- Joint pain
- Rash
- Fever
- Back pain
- Pain in your belly
- Loss of skin color
- Not enough thyroid hormone, so you may feel tired, gain weight, feel cold, or have infrequent or hard stools (hypothyroidism)
- Low levels of salt in the blood that may cause you to feel tired, feel confused, have a headache, have muscle cramps, and/or feel sick to your stomach (hyponatremia)

### UNCOMMON

In 100 people receiving **pembrolizumab**, at least 1 but less than 5 people may have:

- Inflammation of the lungs so you may feel short of breath and cough (pneumonitis)
- Too much thyroid hormone so you may feel anxious, feel angry, have trouble sleeping, feel weak, tremble, sweat, feel tired, have loose and watery stools (hyperthyroidism)
- Infusion reaction, where you may feel dizzy or faint, feel flushed, get a rash, have a fever, feel short of breath, experience a decrease in your blood pressure at the time of receiving your infusion (IV) or just after, or have pain at the site of infusion
- Inflammation of the bowels/gut, which may cause severe pain in your belly with loose or watery stools, and black, tarry, sticky stools or stools with blood or mucus (colitis)
- Inflammation of the skin so you may have peeling of the skin, itchiness, and/or skin redness. The skin inflammation (i.e., peeling, itching and redness) could also be widespread throughout your body. More severe skin reactions may involve the inside of your mouth, the surface of your eye and genital areas, and/or may cause the top layer of your skin to peel from all over your body which can cause severe infection (Severe skin reactions, including Stevens-Johnson syndrome or toxic epidermal necrolysis)

### RARE

In 100 people receiving **pembrolizumab**, less than 1 person may have:

- Inflammation of the nerves that may cause pain, weakness or tingling in your hands and feet, and may spread to your legs, arms and upper body leading to severe muscle weakness and possible temporary paralysis (Guillain-Barré syndrome)
- Inflammation of the muscles, so you may feel week or have pain in your muscles (myositis)
- Inflammation of the pancreas (a gland in your abdomen that controls sugar levels), so you may have severe pain in the top part of your belly that may move to your back, feel sick to your stomach, and have vomiting that gets worse when you eat (pancreatitis)
- Inflammation of the eye so you may have eye redness, blurred vision, sensitivity to light, eye pain, see floaters or have headaches (uveitis)
- Inflammation of the liver that may make you feel sick to your stomach and vomit, feel like not eating, feel tired, have a mild fever, a pain in the right side of your belly, yellow eyes and skin, and dark urine (hepatitis)
- Inflammation of the pituitary gland (a gland in the head), which may cause you to feel sick to your stomach or have headaches, changes in your behavior, double vision, few to no menstrual cycles, weakness, vomiting and dizziness, or fainting (hypophysitis)
- Adrenal glands (glands on top of the kidneys) that may not make enough hormone, which
  could cause tiredness, weight loss, muscle weakness, feeling faint, having joint, muscle,
  and belly aches, nausea, vomiting, loose or watery stools, fever, salt craving, and
  sometimes darkening of the skin like a suntan (adrenal insufficiency)
- Type 1 Diabetes, a condition that can cause too much sugar in your blood, feeling thirstier than usual, frequent urination, and weight loss. You are likely to need regular insulin shots
- Inflammation of the kidney so you may pass less urine or have cloudy or bloody urine, swelling, and low back pain (nephritis)

- Inflammation of the middle layer of your heart wall that may cause your heart to have difficulty pumping blood throughout your body, which can cause chest pain, shortness of breath, and swelling of the legs. You may experience a fast or irregular heartbeat that may cause dizziness or fainting (myocarditis)
- Inflammation of the thyroid gland, an organ that makes and stores thyroid hormones. This condition may lead to change in your heart rate, blood pressure, body temperature, and the rate at which food is converted into energy (thyroiditis)
- A condition that may make you feel weak and tired and may cause drooping of the eyelids, blurred or double vision, difficulty swallowing, slurred speech, weakness in your arms and legs, or difficulty breathing (myasthenic syndrome/myasthenia gravis including exacerbation)
- The formation of small clusters of immune cells (called granulomas) in parts of your body such as your lymph nodes, eyes, skin, or lungs (sarcoidosis)
- Inflammation of the brain with confusion and fever. This may also include: disorientation, memory problems, seizures (fits), changes in personality and behavior, difficulty speaking, weakness or loss of movement in some parts of your body, and loss of consciousness (encephalitis)
- Inflammation of the spinal cord with pain, numbness, tingling, or weakness in the arms or legs, bladder or bowel problems including needing to urinate more frequently, urinary incontinence, difficulty urinating, and constipation (myelitis)
- Inflammation of the blood vessels (vasculitis)
- A condition where the parathyroid glands in the neck do not produce enough parathyroid hormone (PTH) (hypoparathyroidism)

Additionally, since pembrolizumab was first approved in September 2014, the following side effects have been reported by people receiving pembrolizumab. These side effects were voluntarily reported from a group of people of unknown size. It is not possible to estimate the frequency of this side effect:

- Inflammation of the joints which may include joint pain, stiffness and/or swelling (arthritis)
- Severe responses of the immune system that cause the body to attack its own blood cells, spleen, liver, lymph nodes, skin and brain. This may include fever, rash, inflammation of the liver, yellowing of the skin, an enlarged liver and spleen, low blood counts, and enlarged lymph nodes. The nervous system may also be affected and cause confusion, seizures, and even coma (hemophagocytic lymphohistiocytosis)
- Changes in eyesight, eye pain, whitish patches on the skin, and hearing loss (Vogt-Koyanagi-Harada syndrome)
- Inflammation and scarring of the bile ducts (tubes that carry digestive fluid that is made in the liver). This can cause symptoms similar to those seen with inflammation of the liver (hepatitis) such as pain in right side of your belly, yellow eyes and skin, feeling tired, and itching (sclerosing cholangitis).

### **Known Side Effects of Doxorubicin**

### COMMON, SOME MAY BE SERIOUS

In 100 people receiving **doxorubicin**, more than 20 may have:

- Hair loss
- Vomiting
- Red colored urine, saliva, or sweat

### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving **doxorubicin**, from 4 to 20 may have:

- Heart failure or heart attack which may cause shortness of breath, swelling of ankles, cough or tiredness which may occur years after the dose
- Swelling of the body which may cause shortness of breath
- Swelling and redness at the site of the medication injection or area of previous radiation
- Belly pain
- Sores in the mouth, throat or stomach
- Nausea, diarrhea
- Hepatitis which may cause yellow eyes and skin
- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Damage to organs which may cause infection, bleeding, may require transfusions
- Darkening of the nail beds or skin or hands and feet
- Loss of nails

### **RARE. AND SERIOUS**

In 100 people receiving **doxorubicin**, 3 or fewer may have:

- Infection, especially when white blood cell count is low
- Bruising, bleeding
- Severe blood infection
- Cancer of the bone marrow (leukemia) caused by chemotherapy

## **Known Side Effects of Cyclophosphamide**

### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving **cyclophosphamide**, more than 20 may have:

- Hair loss, skin changes, rash, change in nails
- Nausea, vomiting, loss of appetite,
- Pain in belly
- Diarrhea
- · Sores in mouth
- Infection, especially when white blood cell count is low
- Absence of menstrual period which may decrease the ability to have children
- Blood in urine

## OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving **cyclophosphamide**, from 4 to 20 may have:

- Damage to the bone marrow (irreversible) which may cause infection, bleeding, may require transfusions
- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Loss or absence of sperm which may lead to an inability to father children
- · Stuffy nose
- Scarring of the lungs which may cause shortness of breath
- Fluid around the heart

## **RARE, AND SERIOUS**

In 100 people receiving **cyclophosphamide**, 3 or fewer may have:

- Severe skin rash with blisters and peeling which can involve mouth and other parts of the body
- A new cancer including cancer of bone marrow (leukemia) caused by chemotherapy

### **Known Side Effects of Paclitaxel**

### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving **paclitaxel**, more than 20 may have:

- Anemia which may cause tiredness, or may require blood transfusions
- Infection, especially when white blood cell count is low
- Diarrhea
- · Nausea, vomiting
- · Sores in mouth which may cause difficulty swallowing
- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- · Bruising, bleeding
- Pain
- Muscle weakness
- Numbness, tingling or pain of the arms and legs
- Hair loss

### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving **paclitaxel**, from 4 to 20 may have:

- Abnormal heartbeat
- Blood clot which may cause swelling, pain, shortness of breath
- Damage to the lungs which may cause shortness of breath

### **RARE, AND SERIOUS**

In 100 people receiving **paclitaxel**, 3 or fewer may have:

- Heart attack or heart failure which may cause shortness of breath, swelling of ankles, and tiredness
- A tear or a hole in the stomach which may cause belly pain or that may require surgery
- Severe skin rash with blisters and peeling which can involve mouth and other parts of the body

### **Known Side Effects of Nab-Paclitaxel**

### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving **Nab-paclitaxel**, more than 20 may have:

- Swelling of the body
- Infection, especially when white blood cell count is low which can be serious
- Bruising, bleeding
- Anemia, which may cause tiredness, or may require blood transfusions
- Diarrhea, nausea, vomiting, or loss of appetite
- Numbness and tingling of the arms and legs, muscle weakness
- Fever
- Tiredness
- Dehydration
- Hair loss, rash

## OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving **Nab-paclitaxel**, from 4 to 20 may have:

- Heart stops beating
- Mini stroke
- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Abnormal heartbeat
- Blood clot which may cause swelling, pain, shortness of breath
- Damage to the lungs which may cause shortness of breath
- Cloudiness of the eye, visual disturbances
- Pain
- Constipation
- Paralysis, weakness, headache
- Numbness and tingling of the arms and legs
- Hoarseness

### RARE. AND SERIOUS

In 100 people receiving **Nab-paclitaxel**, 3 or fewer may have:

None

## **Known Side Effects of Carboplatin**

Only participants with triple negative breast cancer will receive carboplatin.

### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving **carboplatin**, more than 20 may have:

- Hair loss
- Nausea, vomiting
- Belly pain
- Infection, especially when white blood cell count is low
- Anemia which may cause tiredness, or may require blood transfusions
- Bruising, bleeding

### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving **carboplatin**, from 4 to 20 may have:

- Diarrhea
- Constipation
- Numbness and tingling in fingers and toes
- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Changes in taste
- Changes in vision
- Low levels of magnesium in the blood which could cause muscle weakness and cramping

### **RARE, AND SERIOUS**

In 100 people receiving **carboplatin**, 3 or fewer may have:

- Damage to organs which may cause hearing and balance problems
- Cancer of the bone marrow (leukemia) caused by chemotherapy

### Reproductive Risks

You should not get pregnant, breastfeed, or father a baby while in this study. The treatment used in this study could be damaging to an unborn baby. If you are able to become pregnant, you will need to have a pregnancy test to find out if you can be in the study.

If you participate in this study, you must agree to use a reliable method to prevent pregnancy during all study treatment and for at least 6 months following your last pembrolizumab or decitabine treatment. Check with the study doctor about what methods of preventing pregnancy are acceptable for you.

### **CAN I STOP TAKING PART IN THIS STUDY?**

Yes. You can decide to stop at any time. If you decide to stop for any reason, it is important to let the study doctor know as soon as possible so you can stop safely. If you stop, you can decide whether or not to let the study doctor continue to provide your medical information for the purpose of the study.

The study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study. The study doctor may take you out of the study:

- If your health changes and the study is no longer in your best interest
- If you have serious side effects that require you to stop according to the rules of the study
- If new information becomes available
- If you do not follow the study rules
- If the study is stopped by the sponsor, the FDA, or the institutional review board (IRB), which is a group of people who review the research with the goal of protecting the people who take part in the study

If you withdraw from the study, data that has already been collected about you will remain part of the study database and may not be removed.

### WHAT ARE THE COSTS OF TAKING PART IN THIS STUDY?

Pembrolizumab and decitabine will be supplied at no charge while you take part in this study. It is possible that one or both of these drugs may not continue to be supplied while you are on the study. Although not likely, if this occurs, your study doctor will talk to you about your options.

You will not be charged for any costs related to the needle biopsies to collect tumor samples and to the research using the tumor samples. You will also not be charged for any costs related to the collection and testing of blood samples that are for research purposes.

You and/or your health plan/insurance company will be billed for the standard neoadjuvant chemotherapy, surgery, and all standard costs of treating your cancer, including the cost of tests, procedures, or medicines to manage any side effects.

You will not be paid for taking part in this study.

### WHAT HAPPENS IF I AM INJURED OR HURT BECAUSE I TOOK PART IN THIS STUDY?

If you are injured or hurt as a result of taking part in this study and need medical treatment, please tell your study doctor. Your study doctor or study team will talk with you about your options for medical treatment.

Fees for such treatment may be billed to you or to your health plan/insurance company. Your health insurance company may or may not pay for treatment of injuries or illness as a result of your participation in this study. The study will not pay for medical treatment.

To help decrease the risk of research-related injury or illness, it is very important to follow all study directions.

### WHO WILL SEE MY MEDICAL INFORMATION?

Your privacy is very important to us. The researchers will make every effort to protect it but your information may be given out if required by law. However, the researchers will do their best to make sure that any information that is released will not identify you.

Your research information and your personal identifying information will be kept private through the use of password-protected electronic files, locked research areas, and study identification numbers. Tumor and blood samples will be stored with the same safeguards. When your tumor and blood samples are sent to the laboratory researchers, no information identifying you, such as your name, will be sent. The laboratory researchers will not know who you are. The results of this research may be presented at meetings or in publications, but you will not be identified by name and other personal information will not be used.

There are organizations that may inspect your records. These organizations are required to make sure your information is kept private, unless required by law to provide information. Some of these organizations are:

- Merck & Company, the company providing pembrolizumab for this study
- Virginia Commonwealth University (VCU)
- VCU IRB
- FDA

In the future, the identifiers could be removed from the information and samples you provide for this study. After that removal, your information and samples could be used for new studies without asking for your consent again. Those possible new studies could be done by this study team or other researchers and might involve sequencing all or part of your DNA.

### WHERE CAN I GET MORE INFORMATION?

You may visit the NCI website at <a href="http://cancer.gov/">http://cancer.gov/</a> for more information about studies or general information about cancer. You may also call the NCI Cancer Information Service to get the same information at: 1-800-4-CANCER (1-800-422-6237).

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

### WHO CAN ANSWER MY QUESTIONS ABOUT THIS STUDY?

You can talk to your study doctor or study team about any questions or concerns you have about this study or to report side effects or injuries.

Harry D. Bear, MD, PhD 804-828-9325 Evening/Weekend Doctor 804-828-0951 (Telepage – ask for the hematology/oncology attending doctor on call) Study Team Member 804-628-9238

The Office of Research can answer your general questions or concerns about your rights as a participant in this or any other research. Also, if you would like to speak to a person who does not work directly with your study doctor and the study team or if you cannot reach your study doctor or a member of the study team, you may contact the Office of Research.

Virginia Commonwealth University Office of Research 800 East Leigh Street, Suite 3000, Box 980568, Richmond, VA 23298 804-827-2157; https://research.vcu.edu/human\_research/volunteers.htm

### USE AND DISCLOSURE OF PROTECTED HEALTH INFORMATION

The Health Insurance Portability & Accountability Act (HIPAA) of 1996 provides for the protection of your health information from unauthorized use and disclosure. This section tells you what health information about you may be used and given out in the study and who may give and receive the information. By signing the consent form for this study, you agree that health information that identifies you may be used and disclosed as needed for this research.

### **Authority to Request Protected Health Information**

The following people and/or groups may request your protected health information:

- Sponsor-investigator and research staff
- Study sponsor
- Research collaborators
- VCU IRB
- Data and Safety Monitoring Committee
- Government/health agencies
- Others as required by law

## **Authority to Release Protected Health Information**

The VCU Health System (VCUHS) may release the information identified in this authorization from your medical records and provide this information to:

- Health care providers at the VCUHS
- Sponsor-investigator and research staff
- Research collaborators

- Data coordinators
- VCU IRB
- Data and Safety Monitoring Committee
- Government/health agencies
- Others as required by law

Once your health information has been disclosed to anyone outside of this study, the information may no longer be protected under this authorization.

## Type of Information That May be Released

The following types of information may be used for the conduct of this research:

- Complete health record
- Diagnosis and treatment codes
- Discharge summary
- History and physical exam
- Consultation reports
- Progress notes
- Laboratory test results
- Imaging reports (eg, X-ray reports)
- X-ray films/images
- Information about Hepatitis B, Hepatitis C, and HIV tests
- Complete billing record
- Itemized bill

### **Expiration of This Authorization**

This authorization will expire (end) when the research study is closed or when there is no need to review, analyze, and consider the data generated by the research study, whichever is later.

### Right to Revoke Authorization and Re-disclosure

You may change your mind and revoke (take back) the right to use your protected health information at any time. Even if you revoke this authorization, the researchers may still use or disclose health information they have already collected about you for this study. If you revoke this authorization you may no longer be allowed to participate in the research study. To revoke this authorization, you must write to the sponsor-investigator.

## MY SIGNATURE AGREEING TO TAKE PART IN THIS STUDY

I have been given the opportunity to carefully read this consent form. All of the questions that I wish to raise concerning this study have been answered.

By signing this consent form, I have not given up any of my legal rights or benefits. My signature indicates that I freely consent to participate in this research study. I will receive a copy of the signed consent form.

| Participant Name ( <i>Printed</i> ) | |
|--------------------------------------------------------------|----------|
| Participant Name (Signature) | Date |
| Person Conducting Informed Consent Discussion (Printed Name) | |
| Person Conducting Informed Consent Discussion (Signature) | <br>Date |
| Signature of Investigator ( <i>If different than above</i> ) | <br>Date |